CLINICAL TRIAL: NCT01056198
Title: Comparison of Sharp Surgical Debridement Versus Collagenase Santyl Ointment in the Care of Diabetic Foot Wounds
Brief Title: Santyl vs. Sharp Debridement of Diabetic Foot Wounds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017-101-09-028
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-10

CONDITIONS: Diabetic Foot Ulcers; Foot Wounds
Keywords: Diabetic Foot Ulcers; Diabetic Foot Wounds
MeSH Terms: conditions — Diabetic Foot | interventions — Collagenases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Santyl (Active Comparator): 2 mm Santyl applied once daily
  Interventions: Drug: Santyl
- Control (Sham Comparator): Daily gauze and optional sharp debridement
  Interventions: Procedure: Control

INTERVENTIONS:
Drug: Santyl — 2 mm Santyl applied once daily.
  Arms: Santyl
Procedure: Control — Daily gauze and optional sharp debridement
  Arms: Control

SUMMARY:
This study tests two different approaches to the removal of dead tissue from the surface of a wound.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent document must be read, signed, and dated by the subject or the subject's legally authorized representative before conducting any study procedures or exams. In addition, the informed consent document must be signed and dated by the individual who consents the subject before conducting Visit 1. A photocopy of the signed informed consent document must be provided to the subject, and the original signed document placed in the subject's chart.
* Subjects 18 years of age or older. Subjects may be of either sex and of any race or skin type provided that their skin color, in the opinion of the investigator, will not interfere with the study assessments.
* Willing to make all required study visits.
* Able to follow instructions and perform the dressing changes at home, or, have a caregiver who can perform the dressing changes according to the protocol.
* Willing to use the Darco (orthopedic) shoe off-loading device and insole, if appropriate, starting on the day of screening and running through the follow-up phase.
* A history of Type I or Type II Diabetes Mellitus requiring insulin or oral hypoglycemic medications to normalize blood glucose levels.

A foot wound which is:

* Superficial, involving the full skin thickness but not underlying tissues and is 0.5 cm2 to 10 cm2 in measured surface area at screening visit (not yet debrided)
* Chronic, defined as open for 30 days
* On a neuropathic foot, defined as inability to perceive 10 grams pressure using a Semmes-Weinstein 5.07 or equivalent monofilament in the periwound area
* Adequately perfused, defined as TcPO2 > 40 mmHg; or toe pressure > 40 mmHg, or Doppler waveform consistent with adequate flow in the foot (biphasic or triphasic waveforms) at screening.

  * Acceptable state of health and nutrition with:
* Serum albumin ≥ 2.0 g/dL (20g/L)
* Pre-albumin levels of ≥ 15 mg/dL (0.15g/L).

  * Per Screening lab chemistry† report:
* Alkaline phosphatase <500 U/L
* Alanine aminotransferase (ALT) <200 U/L
* Aspartate aminotransferase (AST) <175 U/L
* Serum total bilirubin <3.0 mg/dL
* Serum blood urea nitrogen (BUN) < 75 mg/dL
* Serum creatinine 4.5 mg/dL
* HbA1c 12%

  * Per Screening lab hematology† report:
* Hemoglobin (Hgb) > 8.0 g/dL
* White blood cells (WBC) > 2.0 109/L
* Absolute neutrophil count > 1.0 109/L
* Platelet count > 50 109/L.

  * Local laboratories will be used, but the ranges for inclusion are set based on Healthpoint Data Management ranges. Refer to Appendix 18.1.2.

Exclusion Criteria:

* Contraindications or hypersensitivity to the use of the study medications or their components (refer to product labels).
* Target wound does not require debridement, or is covered with dry eschar.
* Uncontrolled bleeding disorder.
* Untreated cellulitis extending >2 cm around the target wound, untreated lymphangitic streaking, spread beneath the superficial fascia, deep-tissue abscess, gangrene, or infection of muscle, tendon, joint or bone.
* Infection in a patient with systemic toxicity or metabolic instability (e.g., fever, chills, tachycardia, hypotension, confusion, vomiting, leukocytosis, acidosis, severe hyperglycemia, or azotemia).
* Any of the following:

  * Target wound tunneling per probing and visual assessment
  * Osteomyelitis of the target foot or wound probes to bone
  * Target wound is on the heel
  * Target wound is over a Charcot deformity which cannot be offloaded.
* Diagnosis of chronic granulomatous disease, leukocyte adhesion defects or severe neutropenia
* Treatment with any of the following:

  * Systemic corticosteroids
  * Immunosuppressive agent(s)
  * Chemotherapeutic agent(s)
  * Antiviral agent(s)
  * Platelet-derived growth factor
  * Living skin equivalent
  * Dermal substitute
  * Radiation therapy to the target lower extremity within 30 days prior to signing the informed consent document.
  * Currently on systemic antibiotic therapy
* Any medical condition judged by the Medical Monitor and/or Investigator to cause the study to be detrimental to the subject (specify on the reason for screen failure if this applies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint, Ltd.; Herbert B Slade, MD, Study Director — Healthpoint, Ltd
Locations (9):
- United States (9):
  - Foot Research, Phoenix, Arizona
  - St. Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Advanced Regional Center for Ankle and Foot Care, Altoona, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Paddington Testing Company, Inc., Philadelphia, Pennsylvania
  - Arlington Research Center, Arlington, Texas
  - UNTHSC Fort Worth, Fort Worth, Texas
  - Robert Wunderlich, San Antonio, Texas
  - Providence Health Center, Waco, Texas

REFERENCES:
- [Derived] Tallis A, Motley TA, Wunderlich RP, Dickerson JE Jr, Waycaster C, Slade HB; Collagenase Diabetic Foot Ulcer Study Group. Clinical and economic assessment of diabetic foot ulcer debridement with collagenase: results of a randomized controlled study. Clin Ther. 2013 Nov;35(11):1805-20. doi: 10.1016/j.clinthera.2013.09.013. Epub 2013 Oct 18. PMID 24145042

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4/1/2010 to 8/2/2011 at 7 clinics in the U.S.
Groups:
- Santyl: 2 mm Santyl once daily (QD)
Period: Overall Study
Arm/Group | Santyl | Control
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Santyl | Control | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 9 | 11 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 58.5 (13.3) | 63.5 (9.8) | 61.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Bates-Jensen Wound Assessment Score - Modified (BWAT-m)
Description: The Bates-Jensen Wound Assessment Score was used to collect information about the wound bed appearance in each of 8 categories (sub-scales) each with a possible score of 1 to 5. For each sub-scale intact skin was scored a one (1) while a five (5) would indicate the worst possible rating. All scores were combined to compute a total score for each arm/group, with a score of 8 indicating intact skin (minimum summed score), and a score of 40 indicating the worst possible rating (maximum summed score).
Time Frame: baseline and 28 days
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Santyl | Control
Number analyzed (Participants) | 24 | 24
units on a scale | 15.8 (4.5) | 13.8 (4.8)
Statistical Analysis 1: Comparison: Santyl vs Control; The BWAT-m scores were compared at each of the 4 treatment weeks and at the end of the follow-up using a mixed-effects ANCOVA for the intent-to-treat population. Treatment and treatment week, as well as their interaction, were defined as fixed effects with subject as a random effect. The BWAT-m score at baseline was used as a covariate; Test type: Superiority or Other; p = 0.208, ANCOVA

2. Secondary Outcome: Percent of Wound Area Change From Baseline at End of Treatment
Time Frame: baseline and 28 days
Population: Intent-to-Treat population
Measure: Mean (Standard Error); unit: percentage of baseline wound area
Arm/Group | Santyl | Control
Number analyzed (Participants) | 24 | 24
percentage of baseline wound area | -44.9 (17.0) | 0.8 (57.2)
Statistical Analysis 1: Comparison: Santyl vs Control; Null hypothesis: no differences between the 2 treatments with the alternative of non-zero differences. 48 evaluable subjects is sufficient to detect an effect size of 0.80; Test type: Superiority or Other; p = 0.2737, ANCOVA

3. Secondary Outcome: Percent of Wound Area Change From Baseline at the End of 12 Week Follow-up
Time Frame: baseline and 84 days
Population: Intent-to-Treat population
Measure: Mean (Standard Error); unit: percentage of baseline wound area
Arm/Group | Santyl | Control
Number analyzed (Participants) | 24 | 24
percentage of baseline wound area | -53.8 (17.7) | 8.1 (54.2)
Statistical Analysis 1: Comparison: Santyl vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2741, ANCOVA

4. Post Hoc Outcome: Change From Baseline in Wound Area - Santyl Treatment Group
Description: Wound area at the end of treatment visit compared to the wound area at baseline for each subject
Time Frame: baseline and 28 days
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: square centimeters
Groups:
- Santyl: 2 mm Santyl QD
Arm/Group | Santyl
Number analyzed (Participants) | 24
square centimeters
  Baseline wound area | 3.0 (2.1)
  Wound area at 28 days | 1.8 (2.5)
Statistical Analysis 1: Comparison: Santyl; Paired t-test, 2-sided, alpha = 0.05; Test type: Superiority or Other; p = 0.0164, t-test, 2 sided

5. Post Hoc Outcome: Change From Baseline in Wound Area - Control Group
Description: Wound area at the end of treatment visit compared to the wound area at baseline for each subject
Time Frame: baseline and 28 days
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Control
Number analyzed (Participants) | 24
square centimeters
  Baseline wound area | 2.4 (2.1)
  Wound area at 28 days | 2.3 (4.9)
Statistical Analysis 1: Comparison: Control; Paired t-test, 2-sided, alpha = 0.05; Test type: Superiority or Other; p = 0.9392, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 84 weeks
Arm/Group | Santyl | Control
Serious Adverse Events (participants affected / at risk) | 2/24 | 4/24
Other Adverse Events (participants affected / at risk) | 6/24 | 9/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Santyl (N=24) | Control (N=24)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Peripheral ischemia (Vascular disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Santyl (N=24) | Control (N=24)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Nervous system disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Wound complications (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No